CLINICAL TRIAL: NCT06388538
Title: Conservative vs Surgical (Either Open or Laparoscopic) Approach in the Emergency Management of Acute Diverticulitis WSES 2B: the COLD2B Multicenter, Two-arm Prospective Cohort Study
Brief Title: The COLD2B Multicenter, Two-arm Prospective Cohort Study
Acronym: COLD2B
Status: Not yet recruiting | Type: Observational
Sponsor: Azienda Sanitaria di Firenze (Other)
Responsible Party: Principal Investigator, Alessio Giordano, Principal Investigator, Azienda Sanitaria di Firenze
Other Study IDs: Carlo Bergamini
Record Dates: First submitted 2024-04-20; First posted 2024-04-29 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Acute Diverticulitis
Keywords: COLD2b; acute diverticulitis stage 2B WSES; sigmoid acute diverticulitis; left-side colonic acute diverticulitis
MeSH Terms: interventions — Conservative Treatment; Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with WSES stage 2b acute diverticulitis: Patients with WSES stage 2b acute diverticulitis on the left or sigmoid colon acutely presenting to the emergency departments of the participating centers
  Interventions: Other: Conservative treatment (non-operative treatment); Other: Surgical treatment (operative treatment)

INTERVENTIONS:
Other: Conservative treatment (non-operative treatment) — Conservative treatment consists of medical therapy (see fluid, anti-pain drugs and antibiotics, except for radiologic drainage)
Other: Surgical treatment (operative treatment) — Surgical treatment (operative treatment) is explained as follows:
  1. Open surgery management, i.e. traditional open surgery approach with any kind of technique: either reconstructive (with or without ileal/colonic stoma protection) or non-reconstructive (see Hartman procedure)
  2. Laparoscopic approach, i.e. emergency laparoscopic resection with the characteristics mentioned above

SUMMARY:
Since it is still debated whether 2b acute diverticulitis (AD), according to the World Society of Emergency Surgery (WSES) classification, should be initially treated surgically or conservatively, the COLD2B study has been launched to compare the clinical results of both therapeutic regimens in a multi-institutional cohort of prospectively enrolled patients.

The primary aim of the COLD2B (Conservative vs surgical (either Open or Laparoscopic) approach in the emergency management of acute Diverticulitis WSES 2B) study is to develop a model able to predict the length of hospitalization, comparing the management of WSES 2b AD in the emergency setting (conservative versus surgical approach) (primary endpoint of the first arm of the study).

Moreover, the two groups will be compared regarding mortality and morbidity (secondary end-point).

The second arm of the study will consider the population undergoing surgery, develop a model able to predict the length of hospitalization, and compare the open vs laparoscopic approach (primary end-point), and mortality, morbidity, and surgical outcome indices (secondary end-point).

DETAILED DESCRIPTION:
The COLD2B study is a national, multi-center, prospective observational study of acutely (unplanned and non-elective presentation to hospital for urgent or emergency reasons) presenting patients to the emergency departments of the participating centers with WSES 2b AD (Distant gas - more than 5 cm from inflamed bowel segment).

The study population includes all consecutive adult patients (≥18 years of age) acutely (unplanned and non-elective presentation to hospital for urgent or emergency reasons) presenting at the participating centers with a clinical and radiological diagnosis of WSES 2b AD for 1 year. According to the different management methods, the cohort will be divided into the following categories:

1. Conservatively treated, which will include patients treated with medical therapy (see fluid, anti-pain drugs and antibiotics, except for radiologic drainage) and
2. Surgically resected, which will be devised into the following sub-categories:

2a) Open surgery management, i.e. traditional open surgery approach with any kind of technique: either reconstructive (with or without ileal/colonic stoma protection) or non-reconstructive (see Hartman procedure) 2b) Laparoscopic approach, i.e. emergency laparoscopic resection with the characteristics mentioned above The enrollment period and the overall evaluation will last approximately 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of both sexes, ≥ 18 years old.
2. Patients with abdominal CT scan diagnosis of colonic Acute Diverticulitis classifiable as WSES 2B, i.e..

   1. thickening and other phlegmon signs of the left-sided colonic wall (mostly sigmoid) associated with the inflammatory involvement of the surrounding tissues, plus
   2. presence of air bubbles distant more than 5 cm from the primary colonic inflammatory localization, plus
   3. absence of conspicuous free fluid collection or pelvic abscess.
3. Patients fit for surgery.
4. Patients with colonic diverticulitis on postoperative histological examination.

Exclusion Criteria:

1. Right-sided or transverse diverticulitis
2. Concomitant bowel abscess, perforation, or fistula
3. Radiological drainage
4. Elective procedures.
5. Pregnancy or lactation
6. Patients of both sexes, younger than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by WSES 2b acute diverticulitis actively present at participating hospitals
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Length of hospital stay in the overall population | 1 year
  To develop a predictive model for the length of hospital stay (measured in days) taking into account the treatment received in the overall population

SECONDARY OUTCOMES:
Morbidity rate for both arms | 1 year
  To compare morbidity (i.e. medical problems related to the treatment) for both conservative and surgical arms
Mortality rate for both arms | 1 year
  to compare mortality for both conservative and surgical arms
Surgical complications rate | 1 year
  To compare surgical complications rate for the surgical arms (laparoscopy versus open), measured according to Clavien-Dindo Classification (grade 1 to 5)

CONTACTS AND LOCATIONS:
Locations (4):
- Italy (4):
  - Dipartimento di Medicina di Precisione e Rigenerativa e Area Jonica (DiMePRe-J), Universita' di Bari, Bari
  - Department of Emergency and Acceptance, Emergency Surgery Unit, Azienda Ospedaliero-Universitaria Careggi, Firenze, Italy, Florence
  - Department of Medicine, Surgery and Health Sciences, University of Trieste, Trieste
  - Department of General Surgery, PO di Vittorio Veneto (TV), ULSS2 Marca Trevigiana, Vittorio Veneto

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] undefined
- [Derived] Giordano A, Mastronardi M, Montori G, Anania G, Bergamini C. A focus of therapeutic strategies in acute diverticulitis with distant free air: a systematic review. Updates Surg. 2025 Dec 9. doi: 10.1007/s13304-025-02467-9. Online ahead of print. PMID 41366193
- See also: Hinchey EJ, Schaal PH, Richards MB. Treatment of perforated diverticular disease of the colon. Adv Surg. 1978;12:85-109. — https://pubmed.ncbi.nlm.nih.gov/735943/
- See also: Neff CC, van Sonnenberg E. CT of diverticulitis. Diagnosis and treatment. Radiol Clin N Am. 1989;27:743-52. — https://pubmed.ncbi.nlm.nih.gov/2657852/
- See also: Ambrosetti P, Becker C, Terrier F. Colonic diverticulitis: impact of imaging on surgical management-a prospective study of 542 patients. Eur Radiol. 2002;12:1145-9. — https://pubmed.ncbi.nlm.nih.gov/11976860/
- See also: Kaiser AM, Jiang JK, Lake JP, Ault G, Artinyan A, Gonzalez-Ruiz C, et al. The management of complicated diverticulitis and the role of computed tomography. Am J Gastroenterol. 2005;100:910-7. — https://pubmed.ncbi.nlm.nih.gov/15784040/
- See also: Mora Lopez L, Serra Pla S, Serra-Aracil X, Ballesteros E, Navarro S. Application of a modified Neff classification to patients with uncomplicated diverticulitis. Color Dis. 2013;15:1442-7. — https://pubmed.ncbi.nlm.nih.gov/24192258/
- See also: Sallinen VJ, Leppäniemi AK, Mentula PJ. Staging of acute diverticulitis based on clinical, radiologic, and physiologic parameters. J Trauma Acute Care Surg. 2015;78:543-51. — https://pubmed.ncbi.nlm.nih.gov/25710425/
- See also: Sartelli M, Catena F, Ansaloni L, Coccolini F, Griffiths EA, Abu-Zidan FM, et al. WSES guidelines for the management of acute left sided colonic diverticulitis in the emergency setting. World J Emerg Surg. 2016;11:37. — https://pubmed.ncbi.nlm.nih.gov/27478494/
- See also: Sartelli M, Weber DG, Kluger Y, Ansaloni L, Coccolini F, et al. 2020 update of the WSES guidelines for the management of acute colonic diverticulitis in the emergency setting. World J Emerg Surg. 2020 May 7;15(1):32. — https://pubmed.ncbi.nlm.nih.gov/32381121/
- See also: Francis NK, Sylla P, Abou-Khalil M, et al. EAES and SAGES 2018 consensus conference on acute diverticulitis management: evidence-based recommendations for clinical practice. Surg Endosc. 2019; 33:2726-2741 — https://pubmed.ncbi.nlm.nih.gov/31250244/
- See also: Pavlidis ET, Pavlidis TE. Current Aspects on the Management of Perforated Acute Diverticulitis: A Narrative Review. Cureus. 2022 Aug 26;14(8):e28446. — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC9509703/
- See also: Karentzos A, Ntourakis D, Tsilidis K, Tsoulfas G, Papavramidis T. Hinchey Ia acute diverticulitis with isolated pericolic air on CT imaging; to operate or not? A systematic review. — https://pubmed.ncbi.nlm.nih.gov/33246153/
- See also: Dharmarajan S, Hunt SR, Birnbaum EH, Fleshman JW, Mutch MG. The efficacy of nonoperative management of acute complicated diverticulitis. Dis Colon Rectum. 2011;54:663-71. Int J Surg. 2021;85:1-9 — https://pubmed.ncbi.nlm.nih.gov/21552049/
- See also: Sallinen VJ, Mentula PJ, Leppäniemi AK. Nonoperative management of perforated diverticulitis with extraluminal air is safe and effective in selected patients.. Dis Colon Rectum. 2014;57:875-881 — https://pubmed.ncbi.nlm.nih.gov/24901689/
- See also: Toro A, Mannino M, Reale G, Cappello G, Di Carlo. Primary anastomosis vs Hartmann procedure in acute complicated diverticulitis. Evolution over the last twenty years. Chirurgia (Bucur) 2012;107:598-604. — https://pubmed.ncbi.nlm.nih.gov/23116833/
- See also: Agnes et al Management of acute diverticulitis in Stage 0-IIb: indications and risk factors for failure of conservative treatment in a series of 187 patients. Sci Rep. 2024 Jan 17;14(1):1501 — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC10794215/